CLINICAL TRIAL: NCT01178996
Title: A Phase III, Multicentre, Double Blinded Study In Patients With Chronic Hepatitis C Who Are Non-Responders To Prior Peginterferon Alpha + Ribavirin Therapy Comparing Treatment With Thymosin Alpha 1 + Peginterferon Alpha-2a Plus Ribavirin With Peginterferon Alpha-2a + Ribavirin + Placebo
Brief Title: Thymosin Alpha-1 in Combination With Peg-Interferon Alfa- 2a and Ribavirin for the Therapy of Chronic Hepatitis C Nonresponsive to the Combination of IFN and Ribavirin.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Collaborators: SciClone Pharmaceuticals (Industry)
Responsible Party: Alfonso De Rosa Clinical Research Manager, Sigma-tau SPA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ST1472-DM-03-004; 2004-001277-25 (EudraCT Number)
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Thymalfasin; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thymosin alpha 1 (Experimental): Patients affected by chronic hepatitis C not responding to a course with approved doses of PEGinterferon alpha plus ribavirin therapy (i.e. at least 1.0 mcg/kg PEGinterferon alpha2b, 180 mcg PEGinterferon alfa2a, 800 mg ribavirin).
  Interventions: Biological: Thymosin alpha 1; Drug: Ribavirin; Biological: PEGinterferon alfa2a
- Placebo (Placebo Comparator): Patients affected by chronic hepatitis C not responding to a course with approved doses of PEGinterferon alpha plus ribavirin therapy (i.e. at least 1.0 mcg/kg PEGinterferon alpha2b, 180 mcg PEGinterferon alfa2a, 800 mg ribavirin).
  Interventions: Drug: Ribavirin; Biological: PEGinterferon alfa2a; Drug: Placebo

INTERVENTIONS:
Biological: Thymosin alpha 1 — Thymosin alpha 1 (Zadaxin) 1.6 mg/day, two times weekly in the morning, by subcutaneous injection for 48 weeks.
  Other Names: Zadaxin
  Arms: Thymosin alpha 1
Drug: Ribavirin — Ribavirin 1000 mg (<75 kg) or 1200 mg (>75 kg) daily with food divided in two doses orally for 48 weeks
  Other Names: Copegus
Biological: PEGinterferon alfa2a — 180 mcg, once weekly in the evening, by subcutaneous injection for 48 weeks
  Other Names: Pegasys
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study was to determine safety and efficacy of 48 weeks treatment with Thymosin alpha 1 (Talpha1) in combination with pegylated interferon (PEGIFN) alpha2a and ribavirin (RBV) in adult patients with chronic hepatitis C (CHC) already treated with, and not responding to previous courses of PEGIFN alpha plus RBV combination therapy, in comparison with a concurrent group treated with PEG IFN alpha2a in combination with RBV and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Age 18
3. Presence of HCV RNA measured by quantitative PCR
4. Non responder to previous approved doses of therapy with PEGinterferon alpha plus ribavirin. Patients must have been treated for at least 12 weeks with documented HCV RNA quantitative not showing major of 2 log10 HCV RNA reduction or patients treated for at least 24 weeks with documented HCV RNA qualitative not showing a virological response (viral RNA clearance)
5. Liver biopsy consistent with a diagnosis of chronic hepatitis C or histological cirrhosis. Biopsy will not be required if the patient can produce a biopsy performed within the year preceding the randomization day and was performed at least 6 months after the end of the latter course of therapy
6. Wash-out period of at least 6 months from previous therapy with PEGinterferon alpha plus ribavirin
7. Negative pregnancy test prior (no more than 24 hours) to first study medication dose

Exclusion Criteria:

1. Use of systemic corticosteroids within 6 months of entry
2. More than one previous course of therapy with PEGinterferon alpha plus ribavirin
3. Any other liver disease
4. Decompensated liver disease based on a history of hepatic encephalopathy, bleeding oesophageal varices, or ascites
5. Decompensate or advanced liver cirrhosis (ChildPugh B or C)
6. HIV infection diagnosed by HIV seropositivity and confirmed by Western blot
7. Insulin-dependent Diabetes Mellitus
8. Severe haemoglobinopathy
9. Positive liver and kidney microsomal auto antibodies
10. Positive anti thyroid antibodies
11. Pregnancy as documented by a urine pregnancy test
12. Alcohol or intravenous drug abuse within the previous 1 year
13. Patients who are in poor medical or psychiatric conditions, or who have any non-malignant systemic disease that, in the opinion of the Investigator, would make it unlikely that the patient could complete the study protocol
14. Any indication that the patient would not comply with the conditions of the study protocol
15. Previous treatment with thymosin alpha 1
16. Patients with known hypersensitivity to any PEGinterferon and or ribavirin
17. Patients with a history of severe depression that required either hospitalization or electroshock therapy or depression associated with suicide attempt
18. Simultaneous participation in another investigational drug study or participation in any clinical trial involving investigational drugs within 3 months before study entry
19. Presence of serious pulmonary or cardiovascular disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2004-12; Primary Completion 2008-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Sustained Virological Response (SVR) | Week 72
  The proportion of patients who were HCV RNA negative at the end of observation period.

SECONDARY OUTCOMES:
Sustained Biochemical Response (SBR) | Week 72
  The proportion of patients with normal serum ALT at the end of observation period.
End of Treatment Biochemical Response (EBR) | Week 48
  The proportion of patients with normal serum ALT at the end of treatment period.
End of Treatment Virological Response [EVR] | Week 48
  The proportion of patients who were HCV RNA negative at the end of treatment period.
Safety | During the treatment period (up to 48 weeks) and the follow-up period (up to 24 weeks)
  Safety and tolerability were evaluated by AEs recording, laboratory (hematology and chemistry), ECG, and vital signs evaluations. All laboratory tests were centralized.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Rizzetto, MD, Principal Investigator — Dipartimento Medico Chirurgico delle Malattie dell'Apparato Digerente e della Nutrizione, Azienda Ospedaliera S Giovanni Battista, Corso Bramante 88, Turin, Italy
Locations (9):
- Hôpital Necker, Paris, France
- Universitätsklinikum Tübingen, Tübingen, Germany
- University Hospital of Ioannina, Ioannina, Greece
- Italy (5):
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Policlinico S.Orsola-Malpighi, Bologna
  - Ospedale Cardarelli, Napoli
  - Università Cattolica del Sacro Cuore, Rome
  - Dipartimento Medico Chirurgico delle Malattie dell'Apparato Digerente e della Nutrizione, Azienda Ospedaliera S Giovanni Battista, Turin
- Hospital del Mar, Barcelona, Spain

REFERENCES:
- [Derived] Ciancio A, Andreone P, Kaiser S, Mangia A, Milella M, Sola R, Pol S, Tsianos E, De Rosa A, Camerini R, McBeath R, Rizzetto M. Thymosin alpha-1 with peginterferon alfa-2a/ribavirin for chronic hepatitis C not responsive to IFN/ribavirin: an adjuvant role? J Viral Hepat. 2012 Jan;19 Suppl 1:52-9. doi: 10.1111/j.1365-2893.2011.01524.x. PMID 22233415